CLINICAL TRIAL: NCT05728944
Title: A Multi-Center, Double-Masked Phase 3 Evaluation of the Safety and Efficacy of LNZ101 for the Treatment of Presbyopia
Brief Title: Phase 3 Efficacy Study of LNZ101 for the Treatment of Presbyopia
Acronym: CLARITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LENZ Therapeutics, Inc (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 22-150-0018
Record Dates: First submitted 2023-02-06; First posted 2023-02-15 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Presbyopia; Near Vision; Miosis; Eye Diseases
Keywords: Pharmaceutical Solutions; Opthalmic Solutions; Eye Drops; CLARITY; Presbyopia; Miotic
MeSH Terms: conditions — Presbyopia; Myopia; Miosis; Eye Diseases | interventions — aceclidine

STUDY DESIGN:
Intervention Model Description: A multi-center, double masked, randomized, efficacy and safety study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-masked treatment will be used to reduce potential of bias during data collection and evaluation of clinical endpoints.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Aceclidine + Brimonidine (LNZ101) dosed bilaterally (Experimental): LNZ101: Aceclidine + Brimonidine ophthalmic solution
  Interventions: Drug: Aceclidine+Brimonidine combination ophthalmic solution
- Aceclidine Ophthalmic Solution (LNZ100) dosed bilaterally (Experimental): LNZ100: Aceclidine ophthalmic solution
  Interventions: Drug: Aceclidine
- Vehicle Ophthalmic Solution dosed bilaterally (Experimental): Vehicle ophthalmic solution
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Aceclidine+Brimonidine combination ophthalmic solution — Aceclidine + Brimonidine combination ophthalmic solution
  Other Names: LNZ101
  Arms: Aceclidine + Brimonidine (LNZ101) dosed bilaterally
Drug: Aceclidine — Aceclidine ophthalmic solution
  Other Names: LNZ100
  Arms: Aceclidine Ophthalmic Solution (LNZ100) dosed bilaterally
Drug: Vehicle — Proprietary vehicle ophthalmic solution
  Arms: Vehicle Ophthalmic Solution dosed bilaterally

SUMMARY:
Phase 3 Efficacy Study to evaluate the Safety and Efficacy of LNZ101 for the Treatment of Presbyopia

DETAILED DESCRIPTION:
A Multi-Center, Double-Masked Phase 3 Evaluation of the Safety and Efficacy of LNZ101 for the Treatment of Presbyopia

ELIGIBILITY:
Inclusion Criteria: Subjects MUST:

1. Be able and willing to provide written informed consent and sign a Health Information Portability and Accountability Act (HIPAA) form prior to any study procedure being performed;
2. Be able and willing to follow all instructions and attend all study visits;
3. Be 45-75 years of age of either sex and any race or ethnicity at Visit 1;
4. Have +1.00 to -4.00 diopter (D) of sphere calculated in minus cylinder (so that spherical equivalent (SE) results in myopia no more severe than -4.00 D MRSE) in both eyes determined by manifest refraction documented at Visit 1;
5. Have ≤2.00 D of cylinder (minus cylinder) in both eyes determined by manifest refraction documented at Visit 1;
6. Be presbyopic as determined at Visit 2 baseline

Exclusion Criteria: Subjects must NOT:

1. Be a female of childbearing potential who is currently pregnant, nursing, or planning a pregnancy;
2. Have known contraindications or sensitivity to the use of any of the study medications or their components;
3. Have an active ocular infection at Visit 1 or at Visit 2 (bacterial, viral, or fungal), positive history of an ocular herpetic infection, preauricular lymphadenopathy, or ongoing, active ocular inflammation in either eye;
4. Have moderate or severe dry eye defined as total central corneal fluorescein staining in either eye at Visit 1;
5. Have clinically significant abnormal lens findings including early lens changes during dilated slit-lamp biomicroscopy and fundus exam documented within 3 months of Visit 1 or at Visit 1;

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Efficacy Study To evaluate the safety and efficacy of LNZ101/LNZ100 compared with vehicle for the treatment of Presbyopia. | 3 hours post-treatment in the study eye at Visit 2
  Percentage of subjects who achieve a 3-line or greater improvement from baseline in the study eye.
  compared with vehicle for the treatment of Presbyopia.

CONTACTS AND LOCATIONS:
Overall Officials: Alisyn Facemire, BA, Study Director — LENZ Therapeutics
Locations (13):
- United States (13):
  - Site #209, Dothan, Alabama
  - Site #216, Scottsdale, Arizona
  - Site #214, La Jolla, California
  - Site #203, Newport Beach, California
  - Site #204, Danbury, Connecticut
  - Site #205, Crystal River, Florida
  - Site #211, Louisville, Kentucky
  - Site #208, St Louis, Missouri
  - Site #215, Bozeman, Montana
  - Site #212, West Fargo, North Dakota
  - Site #207, Powell, Ohio
  - Site #213, Eugene, Oregon
  - Site #217, Warwick, Rhode Island

IPD SHARING:
Plan to Share IPD: No